CLINICAL TRIAL: NCT02856997
Title: Chidamide With ICE Regimen for Relapsed/Refractory Peripheral T Cell Lymphoma: A Phase II Clinical Trial
Brief Title: Chidamide With ICE Regimen for Relapsed/Refractory Peripheral T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuankai Shi (Other)
Responsible Party: Sponsor-Investigator, Yuankai Shi, Dr., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAMS 16-059/1138
Record Dates: First submitted 2016-07-24; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide with ICE regimen (Experimental): Drugs:Chidamide and ICE regimen (ifosfamide, Mesna,Carboplatin and etoposide): Chidamide 20mg on d1,4,8,11;ifosfamide 1.2g/ m2，d1-4,ivg during 4 hours; Mesna 0.4g, 0,4,8 hours during Ifosfamide transfusion, ivg, d1-4; Carboplatin AUC=4, d2,ivg; etoposide 65mg/m 2, d1-4, ivg. 3 weeks as 1 course, for 6 courses.
  if the effect is PR or better than PR, go to auto-stem cell transplantation, no further treatment with Chidamide is needed.
  If the effect is PR or better than PR and no auto-stem cell transplantation available,Chidamide 20mg orally, twice every week, till the end of the trial.
  Interventions: Drug: Chidamide with ICE regimen

INTERVENTIONS:
Drug: Chidamide with ICE regimen — Chidamide and ICE regimen, dosage described in arm description
  Other Names: Epidaza，HBI-8000

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Chidamide with ICE regimen in patients with relapsed/refractory Peripheral T Cell lymphoma.

DETAILED DESCRIPTION:
Efficacy of the combined regimen is evaluated primarily by objective remission rate, including complete remission, unverified complete remission and partial remission, also by duration of remission, progression free survival, and overall survival.

Safety is accessed by:

1. The type, incidence, severity of incidents related to the use of the regimen.
2. Laboratory abnormalities, including the type, incidence, severity, relationship with the use of the regimen.
3. Incidence of level 3-4 incidents and laboratory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Peripheral T Cell Lymphoma (PTCL) verified by histopathology/ cytology, according to WHO 2008 classification criteria, including: adult T cell lymphoma or leukemia (human T cell leukemia virus 1 positive); angioimmunoblastic t cell lymphoma; ALK positive anaplastic large cell lymphoma; ALK negative anaplastic large cell lymphoma; non-specified peripheral T cell lymphoma; extra-nodal NK/T cell lymphoma; bowl disease related T cell lymphoma; hepatosplenic T cell lymphoma; subcutaneous panniculitis-like T cell lymphoma; allergic mycosis fungoides.
2. There is at least 1 focus that could be evaluated both by histopathology and cytology (˃1.5cm) according to Cheson criteria.
3. The patients should have had at least 1 course of systemic treatment (including chemo-therapy, stem cell transplantation etc), but did not achieve remission or had relapse after remission.
4. Age18-75 years, male or female;
5. General condition should be ECOG 0-1.
6. Blood routine test: absolute neutrophil count ≥1.5 × 109/L, platelet ≥80 × 109/L, Hb ≥ 90g/L;
7. Expected survival ≥ 3 months;
8. No radiotherapy, chemotherapy, targeted therapy or hemopoietic stem cell transplantation received within 4 weeks prior to enrollment.
9. Willing to sign the written consent.

Exclusion Criteria:

1. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures.
2. QTc elongation with clinical significance ( male˃ 450ms, female˃ 470ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment.
3. Patients who have received organ transplantation.
4. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment.
5. Patients with active hemorrhage.
6. Patients with or with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction.
7. Patients with active infection, or with continuous fever within 14 days prior to enrollment.
8. Had major organ surgery within 6 weeks prior to enrollment.
9. Impaired liver function ( Total bilirubin ˃ 1.5 times of normal maximum, ALT/AST˃ 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST ˃ 5 times of normal maximum), impaired renal function (serum creatinin˃ 1.5 times of normal maximum).
10. Patients with mental disorders or those do not have the ability to consent.
11. Patients with drug abuse, long term alcoholism that may impact the results of the trial.
12. Non-appropriate patients for the trial according to the judgment of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate | through study completion, an average of 30 months

SECONDARY OUTCOMES:
Duration of remission | through study completion, an average of 30 months
progress free survival | through study completion, an average of 30 months
overall survival | through study completion, an average of 30 months
white blood cell count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
red blood cell count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood Hb level | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood platelet count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
vital signs | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum alanine aminotransferase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum aspartate transaminase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum total bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum direct bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum indirect bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum glutamyltranspeptidase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum albumin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum ureal nitrogen level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum creatinin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
fasting blood glucose level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood electrolytes level（K+, Na+，Cl-，Ca2+，Mg2+） | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood LDH level | every 6 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
QTc from ECG | every 6 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months

IPD SHARING:
Plan to Share IPD: Yes
the data of the trial would be open to the public after the trial is finished